CLINICAL TRIAL: NCT05385913
Title: Digital Evaluations and Technologies Enabling Clinical Translation for AD
Acronym: DETECT-AD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: STUDY00023803; 1R56AG074321-01 (NIH)
Record Dates: First submitted 2022-05-16; First posted 2022-05-23 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-10

CONDITIONS: Alzheimer Disease, Early Onset
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood-based laboratory tests include dementia screening laboratories (CBC, chemistry panel, thyroid function, B-12), as well as for exploratory analyses, peripheral blood-based biomarkers related to inflammation (interleukins, CRP), neurodegeneration (NfL, P-tau), vascular risk or injury (HgbA1C, MMP, ICAM, VCAM, VEGF), nutritional health (oxylipins, homocysteine), and genetic risk (apolipoprotein E genotype, and polygenic AD risk or hazard score).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- "Placebo": AB high group; SUVR >1.11
  Interventions: Other: Multivitamin-no intervention
- "Treatment": AB low group; SUVR ≤1.11
  Interventions: Other: Multivitamin-no intervention
- Study Partners: Each participant will also have a stud partner that will be enrolled.

INTERVENTIONS:
Other: Multivitamin-no intervention — No intervention. All participants will be given a multi-vitamin to take for the duration of the study
  Groups: "Placebo"; "Treatment"

SUMMARY:
The DETECT-AD study (stands for "Digital Evaluations and Technologies Enabling Clinical Translation for Alzheimer's Disease") is a new study designed to improve clinical trials for early Alzheimer's disease. DETECT-AD uses specialized home-based digital devices (electronic scale, electronic pill box, under-the-mattress sleep sensor, motion activity sensors, wrist watch activity tracker, driving sensor, and computer software) to see if the devices will improve clinical trial assessments. This 36- month-long study will simulate a clinical trial to determine how well the home system detects clinically meaningful changes. Participants in DETECT will receive a brain scan to assess their risk for developing Alzheimer's Disease.

After the scan, homes will be outfitted with the devices*. Participants will be asked to simply go about their daily routines while data is collected in the background by the digital devices.

The scientists will see if there is a change in the digital assessments in four key areas of life activity:

mobility (walking speed), cognition (computer use), sleep (sleep times), and socialization (time spent out of home). Participants will be asked to take a daily multivitamin as a study 'drug' to mimic clinical trial conditions. Using these methods, the DETECT study will produce outcome measures that reflect real-world everyday function. Establishing the superiority of these novel methods compared to conventional methods (for example, exams in a clinic) will provide a potential new pathway for speeding the development of muchneeded new treatments for Alzheimer's

DETAILED DESCRIPTION:
To achieve this objective, we propose the DETECT-AD (Digital Evaluations and Technologies Enabling Clinical Translation for AD) Study. DETECT-AD is a prospective trial simulation study using a current, extensible, sharable, technology agnostic, and home-based assessment platform that continuously generates DBs and metrics of everyday cognition and function (or Daily Indicators of Active Life - 'DIALS'). The platform also allows for remote capture of conventional clinical assessments as well. A simulated trial study design is used, as there are no current established therapies that will reliably improve meaningful function in stage 1-3 AD10 patients to a degree that one can directly test the sensitivity of DBs or DIALS to treatment mediated change. In short, if there is no change over time in the proposed measure, one would not know if it was a failure of the measure or the treatment. Hence, the use of the simulation paradigm. In this trial, participants with known CNS amyloid (Aβ) status (SUVR-based PET "positive" or "negative") will be enrolled. In the simulation, Aβ "positive" (higher amyloid burden) patients will predictably progress, as if they were receiving placebo; those with less amyloid (Aβ "negative") will have less progression, simulating effective treatment. Primary outcomes will be the change in DBs and DIALS composed of measures in 4 key domains: mobility, cognition, sleep, and socialization. Exploratory analyses of the relationship of the DBs with contemporary imaging (MRI) and blood-based biomarkers related to inflammation, neurodegeneration, vascular risk or injury, and nutritional health will also be conducted.

Impact: Successful completion of this study will provide foundational validated DB and DIALS data improving treatment response readout sensitivity, thus advancing AD clinical trial capability and capacity. The intent is to not only validate a single app or device, but to advance ecologically valid multi-domain assessment, as well as an entire trials-environment specific, DB-facilitated protocol that could be adapted and shared for use by any clinical trial or related study going forward.

ELIGIBILITY:
Inclusion Criteria:

* 1. Sign the informed consent form to enrollment in the protocol 2. Have a study partner available to participate in this study 3. Be 65 or older 4. Living alone or with a cohabitant over age 18 (cohabitant will also be required to consent to the home technology and will be given the option to fully participate in home-based study activities) 5. Be willing to participate in genetic research 6. Ability to have an internet connection at home, financial support supplied by study.

  7. Ability to complete surveys via email on a computer, or cell phone 8. In the opinion of the investigator, be of adequate physical health that participation in the research would not pose a significant risk to the health of the subject 9. Meets criteria for normative (not dementia) cognition, i.e., ≧ Bondi/Jak criteria for MCI 10. If taking an antidepressant, must be on stable dose for at least 12 weeks 11. Study partner is functionally independent and has a MMSE of 24-30, inclusive or Montreal Cognitive Assessment equivalent (adjusted for education, ethnic/racial circumstance).

  12. Participant and study partner are computer literate, defined as able to send and receive an email 13. Household has and uses a desktop, laptop, tablet, or smartphone 14. Lives in a residence composed of at least a living space and bathroom

Exclusion Criteria:

* 1. Significant neurologic disease such as AD, multi-infarct dementia, Parkinson's disease, normal pressure hydrocephalus, brain tumor, cortical infarct on MRI, or a history of significant head trauma with subsequent persistent neurologic deficits.

  2. Major psychiatric disorder such as major depression, bipolar disorder (DSM-IV criteria), or history of schizophrenia (DSM-IV). Psychotic features, agitation or behavioral problems within the last 3 months which could lead to difficulty complying with the protocol.

  3. History of alcohol or substance abuse or dependence within the past 2 years (DSM-IV criteria).

  4. Uncontrolled medical conditions precluding completion of the study, e.g., late-stage cancers.

  5. Cannot undergo neuroimaging procedures (e.g., claustrophobia, metallic implants) 6. More than two people live in the participant's residence (overnight visitors are acceptable).

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: older adults living independenlty and/or with a partner; cognitively healthy and/or MCI; ages 65 or older
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Progression of DB's | 36 months
  Determine rates of progression of DBs (of mobility, cognition, sleep, and social engagement) individually and as an aggregate metric (the DIALS) in stage 1-3 Aβ (+) vs. Aβ (-) participants. Early base rates (first months of monitoring) of progression, and then, longitudinal change will be established.
Utility of DB's | 36 months
  Establish the utility of these DBs compared to conventional measures used in trials (i.e., CDR-SoB, ADCS-PACC) by providing meaningful change readout earlier than conventional measures.

SECONDARY OUTCOMES:
Investigate exploratory Aims | 36 months
  Investigate exploratory aims examining several high-value featurse of these DB's for application in trials and clinical studies: Correlate DBs and DIALS with conventional imaging and blood-based biomarkers; inflammation (interleukins, CRP), neurodegeneration (P-tau 181 and 231, NfL), vascular risk or injury (HbgA1C, MMP 1/2/3/9, ICAM, VCAM, VEGF) and nutritional health (oxylipins, homocysteine)
Change over time | 36 months
  Determine the change overtime of embedded cognitive clocks (time to complete regular weekly online report queries and monthly cognitive tests)
Establish adverse event fluctuations over time | 36 months
  (mood, illness, pain, ER, doctor, hospital visits, falls and injury, non-study medication changes) via weekly remote assessments
assess study partner | 36 months
  assess the study partners DB's change relative to the simulated treated study participant (mobility, sleep, social engagement)

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided